CLINICAL TRIAL: NCT00674089
Title: Evaluation of the Effectiveness of Vitamin A Supplementation (VAS) as Part of a Neonatal Post Partum Care Package in Rural Pakistan
Brief Title: Newborn Vitamin A (VA) Supplementation Pilot Project, Pakistan
Acronym: VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: John Snow, Inc. (Industry); Pakistan Ministry of Health (Other Government); Save the Children (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Prof. Zulfiqar A Bhutta, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 586-Ped/ERC-06
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2010-10

CONDITIONS: Vitamin A Deficiency
Keywords: IMR; Newborn Mortality; Vitamin A Effectiveness; Premature Mortality; Mortality
MeSH Terms: conditions — Vitamin A Deficiency | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Routine Post-partum Care and Vitamin A supplementation (50,000 IU) to the Newborn
  Interventions: Dietary Supplement: Vitamin A
- 2 (Placebo Comparator): Routine Post-partum Care with Placebo to the Newborn
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin A — Vitamin A 50,000 IU
  Arms: 1
Dietary Supplement: Placebo — Vitamin A Placebo
  Arms: 2

SUMMARY:
Vitamin A is an essential micronutrient for the normal functioning of the visual system, growth and development, immunity and reproduction. Its deficiency causes anemia, growth retardation and xerophthalmia. Vitamin A deficiency also increases the incidence and/or severity of infectious episodes and affects child survival. Reduced child survival is the most severe and potentially the most widespread consequence of Vitamin A deficiency. Improvement in vitamin A status is now regarded as one of the most cost effective preventive measures for the reduction of child mortality and morbidity.

Over the past decade several studies have examined the effect of vitamin A on reducing mortality among children aged ≥6months at the time of intervention. Impact of vitamin A supplementation can significantly reduce total mortality but it is only established through supplementation programs in children age 6 months or older. It was assumed that breast milk protects infants from vitamin A deficiency, but recent evidence has challenged this. Infants born with low stores of vitamin A and if the mother breast milk has a low concentration of vitamin A, as found in developing countries, the infants might be unable to meet their daily requirements and improve body reserves. There is association between mortality and degree of vitamin A deficiency, greater the degree of deficiency, higher the mortality.

The role of vitamin A in child survival is now well established and over 60 countries have vitamin A supplementation programs nationally. However, most are still using vitamin A supplements in the second half of infancy, even though over 75% of all under 5 deaths take place in the first 6 months of life. If neonatal vitamin A supplementation can be found to be effective and a service delivery mechanism also found, this will represent a major advance in reaching the MDG 4 targets. This is thus persuasive reason to explore this particular preventive strategy, especially in terms of packaging with other postnatal care activities. However, given that in some instances it has been difficult to disentangle the effect of vitamin A dosing from concomitant vaccinations such as BCG, the current evidence needs further evaluation in effectiveness settings. We propose to evaluate the effectiveness of early neonatal vitamin A administration (single dose 50,000 units) to the newborn to see its effect on infant mortality less than 6 months of age as part of postnatal package through National Program.

Government has launched the National Program for Family Planning and Primary Health Care since April 1994. Primarily it is being implemented in the community through Lady Health Workers (LHWs) of the National Program.

The LHWs are females, with a minimum of eight years of education, residents of the locality in which they are working. The Programme is being currently implemented in all the districts throughout the country and 93,000 LHWs are working covering primarily women and children of the rural population. These LHWs deliver services related to family planning, maternal and child health, immunization, nutrition and treatment of minor ailments to her average registered population of 100-150 households or ~1000 population. Over 3,000 Supervisors have been recruited and trained to supervise the work of LHWs.

DETAILED DESCRIPTION:
Goal:

To reduce the infant mortality rate in rural Pakistan through evidence based interventions.

Aim:

To evaluate the impact of a community-based neonatal Vitamin A supplementation program on the morbidity and mortality in newborns and young infants (1-6 months of age) when administered at community level

Primary objectives:

1. To evaluate the effectiveness of a single dose 50,000 IU of vitamin A supplementation to newborn infants within 48 hours after birth in rural Punjab and Sindh in reducing mortality (<6 months of age) by ≥ 25%.
2. To evaluate the feasibility of neonatal vitamin A dosing when administered by LHW as part of postnatal care package

Methodology:

Study Design: Community based, cluster randomized, double blinded, placebo control trial

Sample size estimation:

Assuming average infant mortality rate 40 per thousand live births in the proposed clusters without intervention (range 30-50/1000 live births), and a targeted 25% reduction in mortality in first six months of life, (5% significance level and 80% power) our estimates indicate that the trial will require total 360 clusters [180 in each arm]. The average population size and birth rate per LHW are 1000 and 30 respectively Study Site: Districts Sukkhur and Jehlum. Both the districts, represent a typical mix of peri-urban and rural, multiethnic population of Pakistan. Although a public health care infrastructure exists, it is notable that almost 60% of the population seeks care from private health sector. Current rates of immunizations are poor (approximately 60%) and largely population is illiterate.

ELIGIBILITY:
Inclusion Criteria:

* Live born infants from all pregnancies within participating villages will be eligible for enrollment in this study.

Exclusion Criteria:

* Child born with congenital malformation
* Serious birth injury
* Neonates with birth asphyxia and serious infections
* Gestational age less than 32 weeks
* Birth weight less than 1500 gms
* Refusal by parents to participate

Max Age: 15 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7400 (Actual)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome is reduction in Infant Mortality less than six months of age | 2 years

SECONDARY OUTCOMES:
Secondary outcomes includes reduction in the incidence of diarrhea, ARI and Sepsis | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Project Office, Sukkur, Sindh, Pakistan

REFERENCES:
- [Derived] Soofi S, Ariff S, Sadiq K, Habib A, Bhatti Z, Ahmad I, Hussain M, Ali N, Cousens S, Bhutta ZA. Evaluation of the uptake and impact of neonatal vitamin A supplementation delivered through the Lady Health Worker programme on neonatal and infant morbidity and mortality in rural Pakistan: an effectiveness trial. Arch Dis Child. 2017 Mar;102(3):216-223. doi: 10.1136/archdischild-2016-310542. Epub 2016 Jun 28. PMID 27471856